CLINICAL TRIAL: NCT07004530
Title: Magnetically Controlled Capsule Endoscopy vs Esophago-gastro-Duodenoscopy as The Initial Investigation for Anaemia in Patients With Acute Coronary Syndrome (the MCCE vs EGD Trial) - a Single Centre Randomized Study
Brief Title: the MCCE vs EGD Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, GuangMing Tan, Assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024.237
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Anaemia; Acute Coronary Syndrome
Keywords: Capsule Endoscopy; Esophago-gastro-Duodenoscopy
MeSH Terms: conditions — Anemia; Acute Coronary Syndrome | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients meeting eligibility criteria will be randomized by one of the research team staff via sealed envelopes with computer generated randomization number to one of the two study arms (0 for EGD, 1 for CE) in a 1:1 ratio, according to a central randomization scheme. Due to the nature of the interventions, researchers and patients are not blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCCE-first arm (Experimental): MCCE will be performed for individuals randomized to MCCE arm within the same hospitalization of ACS diagnosis. The MCCE used in this study is the magnetically controlled capsule endoscopy (MCE, AnPx USA) which is a capsule measuring 28x12mm, and contains a permanent magnet inside its dome. Images are captured and recorded at 2 frames/s. Before the MCCE procedure, subjects will be fasted for 8 hours. Capsule will be swallowed with 10ml of clear liquid. During the MCCE examination, subjects will be asked to drink 500 to 1000ml water on demand. Once inside the stomach, the capsule will be navigated via an external magnetic guidance system to obtain a full view of the stomach. After the gastric examination, the subject wears a portable image recorder for images of duodenum and the rest of the small bowel for about 4 hours
  Interventions: Procedure: Magnetically Controlled Capsule Endoscopy (MCCE)
- EGD-first arm (Experimental): Conventional EGD with intravenous sedation will be performed for individuals randomized to EGD arm within the same hospitalization of ACS diagnosis by an experienced endoscopist. Similar MLD and Forest ulcer grading will be applied as in MCCE arm. Endoscopic therapeutic procedures will be performed at endoscopist's discretion.
  Interventions: Procedure: Esophageal-gastro-Duodenoscopy (EGD)

INTERVENTIONS:
Procedure: Magnetically Controlled Capsule Endoscopy (MCCE) — . The MCCE used in this study is the magnetically controlled capsule endoscopy (MCE, AnPx USA) which is a capsule measuring 28x12mm, and contains a permanent magnet inside its dome. Images are captured and recorded at 2 frames/s
  Arms: MCCE-first arm
Procedure: Esophageal-gastro-Duodenoscopy (EGD) — Esophageal-gastro-Duodenoscopy (EGD) is commonly performed to look for source of bleeding in patients with anaemia. However, from our own analysis and from retrospective studies of EGD in patients with ACS, EGD finding was normal or non-significant in 20-80% patients14-16. Moreover, EGD was associated with non-negligible periprocedural risks in patients with ACS, including death directly attributed to EGD (9.1%; 95% CI 7.6-10.9%), hypotension (24.1%; 95% CI 17.0-32.9%), arrhythmias (8.3%; 95% CI 4.5-15.1%) and recurrent ACS (6.5%; 95% CI 3.2-12.8%)
  Arms: EGD-first arm

SUMMARY:
Anaemia is common in patients with acute coronary syndrome (ACS) and is associated with significant recurrent bleeding risk and major adverse cardiovascular event (MACE). Esophageal-gastro-Duodenoscopy (EGD) is commonly used as an initial investigation for anaemia but is often non-diagnostic. Magnetically Controlled Capsule Endoscopy (MCCE) being less invasive and with comparable diagnostic accuracy as EGD, might be used as an alternative initial investigation for anaemia in patients with ACS.

DETAILED DESCRIPTION:
Anaemia is common in patients with acute coronary syndrome (ACS) and is associated with significant recurrent bleeding risk and major adverse cardiovascular event (MACE). Esophageal-gastro-Duodenoscopy (EGD) is commonly used as an initial investigation for anaemia but is often non-diagnostic. Magnetically Controlled Capsule Endoscopy (MCCE) being less invasive and with comparable diagnostic accuracy as EGD, might be used as an alternative initial investigation for anaemia in patients with ACS.

ELIGIBILITY:
Inclusion Criteria:

subjects are patients older than 18 years old with:

1. the diagnosis of ACS as defined by symptoms of chest pain or shortness-of-breath, abnormal electrocardiogram and positive enzyme, requiring coronary intervention
2. new-onset anaemia as defined by Hb<11 g/dL on admission blood taking

Exclusion Criteria:

1. History of active haematological disease including hemoglobinopathies such as thalassemia, Myelodysplastic syndromes, haematological malignancy, aplastic anaemia, or autoimmune haemolytic anaemia.
2. Patients with known active gastrointestinal malignancy.
3. Contraindications for CE: suspected or known gastrointestinal obstruction, stenosis, fistula, diverticula, presence of gastrointestinal obstruction symptoms such as pain or dysphagia; inoperative conditions or refusal to undergo abdominal surgery if required; history of laparotomy, gastric or bowel surgery; presence of metallic implants that is not MRI conditional.
4. Contraindications for EGD: Possible gastrointestinal perforation, medically unstable patients, patient with known pharyngeal diverticulum, and patients with recent head and neck trauma.
5. Inability to take 1-month DAPT such as non-deferrable surgery within 1 months, severe allergy or hypersensitivity reaction to aspirin or P2Y12 inhibitors, or patients in whom 1 months DAPT is not indicated.
6. Patients whose life-expectancy is less than 6 months.
7. Patients who are pregnant or lactating.
8. Patients who are unable to give informed consent.
9. Patients who are in active heart failure or fluid-overload state.
10. Patients who have chronic renal failure as defined by estimated glomerular filtration rate <15 ml/min/1.73m2.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-09-24 (Estimated); Primary Completion 2027-09-24 (Estimated); Study Completion 2027-11-24 (Estimated)

PRIMARY OUTCOMES:
the occurrence of recurrent bleeding | baseline, 30 days
  A bleeding event will be defined according to international consensus by the occurrence of any of the followings: 1) overt bleeding of gastroduodenal origin including fresh hematemesis, bloody nasogastric aspiration, melena after normalization of stool colour, or haematochezia after normalization of stool colour, or 2) bleeding of presumed occult gastrointestinal origin with a documented reduction in haemoglobin concentration of ≥2 g/dl or reduction in the haematocrit by 10% or more from the baseline.

SECONDARY OUTCOMES:
Need for any transfusion | baseline, 30 days
  Need for any transfusion
Any bleeding by Thrombolysis in Myocardial Infarction (TIMI), Bleeding Academic Research Consortium (BARC) and GUSTO definitions | baseline, 30 days
  TIMI flow grade is a method used to assess coronary artery blood flow during and after thrombolytic therapy in patients with acute myocardial infarction. It's a standardized way to grade the degree of reperfusion, ranging from complete occlusion (Grade 0) to complete perfusion (Grade 3).
  BARC:
  Type 1: Minimal bleeding, not actionable. Type 2: Clinically evident but minor; requires treatment. Type 3: Significant bleeding, divided into 3A (moderate, requires transfusion), 3B (major, may need surgery), and 3C (critical, such as intracranial bleeding). Type 4: Bleeding related to CABG procedures.
Change in Major adverse cardiac events | baseline, 30 days
  MACE as defined by death of cardiovascular origin, non-fatal myocardial infarction, non-fatal stroke, or clinically driven target vessel revascularization.
Any adverse events and complications from MCCE and/or from EGD | baseline, 30 days
  Any adverse events and complications from MCCE and/or from EGD

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong